CLINICAL TRIAL: NCT06725446
Title: Correlation Between Symptoms and Hystroscopic Findings in Patients with Uterine Niche: Cross-sectional Study.
Brief Title: Uterine Niche Symptoms and US and Hystroscopic Findings
Acronym: Uterine niche
Status: Active, not recruiting | Type: Observational
Sponsor: Amira Hasan Abdelhady (Other)
Responsible Party: Sponsor-Investigator, Amira Hasan Abdelhady, Principal investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Niche symptoms and findings
Record Dates: First submitted 2024-12-03; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Uterine Niche

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | US Export: No

SUMMARY:
correlation between clinical ,soonographic and hysteroscopic findings in patients with uterine niche

ELIGIBILITY:
Inclusion Criteria:

* patient with uterine niche previous cs

Exclusion Criteria:

abnormal uterine bleeding

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: patients with abnormal uterine bleeding previous cs
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
uterine niche symptoms and Hystroscopic and US findings | 2023-2025
  The correlation between uterine niche symptoms and the hystroscopic and sonographic findingd

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt